CLINICAL TRIAL: NCT02541461
Title: Changes in Lipid Indices and Body Composition One Year After Laparoscopic Gastrectomy: a Prospective Study
Brief Title: Body Composition After Laparoscopic Gastrectomy for Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University Seoul Hospital (Other)
Responsible Party: Principal Investigator, Ji Young Kim, Clinical Professor, Hanyang University Seoul Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-04-026-002
Record Dates: First submitted 2015-09-01; First posted 2015-09-04 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Gastric Cancer; Benign Gastric Tumor
Keywords: Body composition measurement; Lipid profile; Weight loss; Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-Obese (Other): Patients who underwent laparoscopic gastrectomy and with BMI < 25 kg/m2
  Interventions: Procedure: Laparoscopic gastrectomy
- Obese (Other): Patients who underwent laparoscopic gastrectomy and with BMI ≥ 25 kg/m2
  Interventions: Procedure: Laparoscopic gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic gastrectomy — (1) Wedge resection, subtotal or total gastrectomy with or without lymph node dissection; (2) R0 resection; (3) Laparoscopic gastrectomy; (4) Gastroduodenal anastomosis or duodenal bypass, including Roux-en-Y or gastrojejunostomy

SUMMARY:
Nutritional status including changes of body composition is one of the most important clinical determinants of outcome after gastrectomy for gastric cancer. Various type of gastric operations are widely used with favorable outcome in South Korea. It was reported that several advantages of laparoscopic gastrectomy are the prevention of overt weight loss and enhanced recovery of muscle mass at 6 months after surgery. But there have been no longitudinal studies evaluating changes in the body composition according to the different type of anastomosis of laparoscopic gastrectomy.

The purpose of this prospective study was to investigate changes in lipid indices associated with whole body composition during 1 year of follow-up after laparoscopic gastrectomy. Gastrectomy resulted in improved lipid indices and a reduction in body weight, fat and LBM. The HDL-Csignificantly increased in the non-obese group for 1 year after gastrectomy and the reduction of TG level was positively correlated with fat, especially with trunk fat.

DETAILED DESCRIPTION:
* All patients will undergo a laparoscopic gastrectomy for their gastric cancer (proved to be stage I or II) or benign gastric neoplasm by preoperative screening diagnostic procedure. They will receive laparoscopic gastrectomy as follows: (1) wedge resection, subtotal or total gastrectomy with or without lymph node dissection; (2) R0 resection; (3) laparoscopic gastrectomy; (4 gastroduodenal anastomosis or duodenal bypass, including Roux-en-Y or gastrojejunostomy.
* Pre-operative, 6 and 12 months post-operative body composition measurement will be performed on each patient. The whole body composition measurement will be assessed by Hologic 4500/A dual energy X-ray absorptiometry system. The software performs calculations of the differential attenuations of the two photon energies and present data of percentage of fat, fat mass (g), lean mass (g), bone mineral content (g), bone mineral density (g/cm2), and total mass (g).
* Laboratory analysis - There is a battery of labs that are ordered in both the pre-operative, 6 and 12 months post-operative time frame. These labs are ordered independent of the patient's participation in the study. These labs are ordered to evaluate and to assist management of the patient's medical comorbidities as well as to assess for adequate nutritional intake and balance.
* Queries on nutritional intake and exercise will be made at each post-operative appointment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with gastric cancer or benign gastric neoplasm planning gastric operation
* Stage I and II patients by preoperative screening

Exclusion Criteria:

* Distant metastasis
* Severe comorbidity
* Malnourished state
* Inability of access to enteral feeding

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in body composition (changes in lean tissue mass and fatty tissue mass Using DEXA machine produced by Hologic) | pre-surgery, 6 and 12 months post-surgery
  Using DEXA machine produced by Hologic (QDR 4500), changes in lean tissue mass and fatty tissue mass following gastric operation assessed

SECONDARY OUTCOMES:
Changes in lipid profile | pre-surgery, 6 and 12 months post-surgery
  Using laboratory analysis, changes in the lipid profiles (total cholesterol (TC), triglyceride (TG), LDL-C and HDL-C) following gastric operation assessed

CONTACTS AND LOCATIONS:
Overall Officials: Yun Young Choi, MD, PhD, Principal Investigator — Hanyang University Seoul Hospital
Locations (1):
- Hanyang University Seoul Hospital, Seoul, South Korea

REFERENCES:
- [Background] Song J, Lee HJ, Cho GS, Han SU, Kim MC, Ryu SW, Kim W, Song KY, Kim HH, Hyung WJ; Korean Laparoscopic Gastrointestinal Surgery Study (KLASS) Group. Recurrence following laparoscopy-assisted gastrectomy for gastric cancer: a multicenter retrospective analysis of 1,417 patients. Ann Surg Oncol. 2010 Jul;17(7):1777-86. doi: 10.1245/s10434-010-0932-4. Epub 2010 Feb 12. PMID 20151217
- [Background] Kitano S, Iso Y, Moriyama M, Sugimachi K. Laparoscopy-assisted Billroth I gastrectomy. Surg Laparosc Endosc. 1994 Apr;4(2):146-8. PMID 8180768
- [Background] Lee HJ, Kim HH, Kim MC, Ryu SY, Kim W, Song KY, Cho GS, Han SU, Hyung WJ, Ryu SW; Korean Laparoscopic Gastrointestinal Surgery Study Group. The impact of a high body mass index on laparoscopy assisted gastrectomy for gastric cancer. Surg Endosc. 2009 Nov;23(11):2473-9. doi: 10.1007/s00464-009-0419-1. Epub 2009 Apr 3. PMID 19343439
- [Background] Kim MC, Kim W, Kim HH, Ryu SW, Ryu SY, Song KY, Lee HJ, Cho GS, Han SU, Hyung WJ; Korean Laparoscopic Gastrointestinal Surgery Study (KLASS) Group. Risk factors associated with complication following laparoscopy-assisted gastrectomy for gastric cancer: a large-scale korean multicenter study. Ann Surg Oncol. 2008 Oct;15(10):2692-700. doi: 10.1245/s10434-008-0075-z. Epub 2008 Jul 29. PMID 18663532
- [Background] Kim HH, Hyung WJ, Cho GS, Kim MC, Han SU, Kim W, Ryu SW, Lee HJ, Song KY. Morbidity and mortality of laparoscopic gastrectomy versus open gastrectomy for gastric cancer: an interim report--a phase III multicenter, prospective, randomized Trial (KLASS Trial). Ann Surg. 2010 Mar;251(3):417-20. doi: 10.1097/SLA.0b013e3181cc8f6b. PMID 20160637
- [Background] Liedman B, Svedlund J, Sullivan M, Larsson L, Lundell L. Symptom control may improve food intake, body composition, and aspects of quality of life after gastrectomy in cancer patients. Dig Dis Sci. 2001 Dec;46(12):2673-80. doi: 10.1023/a:1012719211349. PMID 11768259
- [Background] Kiyama T, Mizutani T, Okuda T, Fujita I, Tokunaga A, Tajiri T, Barbul A. Postoperative changes in body composition after gastrectomy. J Gastrointest Surg. 2005 Mar;9(3):313-9. doi: 10.1016/j.gassur.2004.11.008. PMID 15749590
- [Background] Abdiev S, Kodera Y, Fujiwara M, Koike M, Nakayama G, Ohashi N, Tanaka C, Sakamoto J, Nakao A. Nutritional recovery after open and laparoscopic gastrectomies. Gastric Cancer. 2011 Jun;14(2):144-9. doi: 10.1007/s10120-011-0021-9. Epub 2011 Feb 16. PMID 21327442
- [Background] Aoyama T, Yoshikawa T, Hayashi T, Hasegawa S, Tsuchida K, Yamada T, Cho H, Ogata T, Fujikawa H, Yukawa N, Oshima T, Rino Y, Masuda M. Randomized comparison of surgical stress and the nutritional status between laparoscopy-assisted and open distal gastrectomy for gastric cancer. Ann Surg Oncol. 2014 Jun;21(6):1983-90. doi: 10.1245/s10434-014-3509-9. Epub 2014 Feb 6. PMID 24499830
- [Background] Jeon TY, Lee S, Kim HH, Kim YJ, Lee JG, Jeong DW, Kim YJ. Long-term changes in gut hormones, appetite and food intake 1 year after subtotal gastrectomy with normal body weight. Eur J Clin Nutr. 2010 Aug;64(8):826-31. doi: 10.1038/ejcn.2010.83. Epub 2010 May 19. PMID 20485300
- [Background] Liedman B, Henningsson A, Mellstrom D, Lundell L. Changes in bone metabolism and body composition after total gastrectomy: results of a longitudinal study. Dig Dis Sci. 2000 Apr;45(4):819-24. doi: 10.1023/a:1005420416192. PMID 10759255